CLINICAL TRIAL: NCT00086671
Title: A 24-Week, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled, Dose Finding, Safety, Tolerability, and Efficacy Study of the Human Anti-IL-12 Antibody ABT-874 in Subjects With Multiple Sclerosis With a 24-Week Double-Blind, Active Extension Phase
Brief Title: Safety and Effectiveness of Two Doses of ABT-874 as Compared to Placebo in Subjects With Multiple Sclerosis (MS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: M03-654
Record Dates: First submitted 2004-07-07; First posted 2004-07-09 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2013-01

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ABT-874 200 mg weekly (Experimental)
  Interventions: Drug: ABT-874/Human monoclonal antibody against IL-12
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- ABT 874 QOW (Experimental)
  Interventions: Drug: ABT-874/Human monoclonal antibody against IL-12

INTERVENTIONS:
Drug: ABT-874/Human monoclonal antibody against IL-12
  Arms: ABT 874 QOW; ABT-874 200 mg weekly
Drug: Placebo
  Arms: Placebo

SUMMARY:
The objective of the trial is to study the safety and effectiveness of ABT-874 administered weekly or every other week in patients with relapsing remitting and secondary progressive multiple sclerosis as compared to placebo. Effectiveness will be measured based on MRI scans done periodically throughout the study.

DETAILED DESCRIPTION:
This study was done in subjects with relapsing remitting MS or secondary progressive MS with the objective of assessing the safety and efficacy of 200 mg of ABT-874 weekly or QOW versus placebo. There were 3 phases to the study, 24 week double blind followed by 24 weeks of an active extension, followed by 48 weeks of double blind active extension. The trial was discontinued by Abbott in Aug 2006.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 55 years
* Diagnosis of active relapse within 12 months of screening.
* At least one relapse within 12 months of screening.
* Must be able to walk at least 65 feet with or without assistance
* Off Copaxone or interferon therapy for two months prior to screening
* Able and willing to learn to self-administer weekly injections, or have a designee who will administer study medication
* Female participants must use contraceptives while on study drug

Exclusion Criteria:

* Primary progressive multiple sclerosis (PPMS)
* Immunosuppressive therapy (such as azathioprine, methotrexate (MTX), but excluding corticosteroids) within six months of randomization. Subjects with previous treatment with cyclophosphamide, total lymphoid irradiation, mitoxantrone, cladribine, or bone marrow transplantation, regardless of duration, will be excluded from participation in this study
* Systemic corticosteroid therapy within four weeks prior to the first screening Magnetic Resonance Imaging (MRI)
* Participation in any clinical study, whether or not it involves an investigational drug within three months prior to the screening visit
* Use of any investigational drug with disease-modifying potential for the treatment of multiple sclerosis (MS) within six months of randomization (prior use of investigational agents for the symptomatic treatment of MS, e.g., 4-aminopyridine (4-AP), may be allowed following discussion with medical monitor
* Concomitant statin use in doses exceeding the manufacturers' maximum recommended daily dosages for treatment of hypercholesterolemia or as part of an MS disease-modifying protocol
* Infection or risk factors for severe infections
* Excessive immunosuppression or other factors associated with it, including human immunodeficiency virus (HIV) infection
* Severe, recurrent, or persistent infections [such as Hepatitis B or C, or borreliosis or recurrent urinary tract infection (UTI) (> 3 UTIs requiring antibiotic treatment per year) or recurrent pneumonia (> 2 pneumonias requiring antibiotic treatment per year) or infected decubitus ulcers]
* Evidence of current inactive tuberculosis (TB) infection; recent exposure to mycobacterium tuberculosis (converters to a positive purified protein derivative [PPD]). Subjects with a positive PPD or a chest X-ray suggestive of prior TB infection will be excluded
* Active tuberculosis disease
* Active chronic Lyme disease
* Active syphilis
* Any other significant infection requiring hospitalization or intravenous (IV) antibiotics in the month prior to Screening; or
* Infection requiring treatment with antibiotics in the two weeks prior to Screening.
* Any of the following risk factors for development of malignancy:

  * History of lymphoma or leukemia
  * Cutaneous squamous-cell or basal cell carcinoma (EXCEPT if treated more that two years prior to Screening with evidence of recurrence or residual disease)
  * Other malignancy (EXCEPT if treated more than five years prior to Screening without evidence of recurrence or residual disease) or
  * Disease associated with an increased risk of malignancy (such as familial polyposis).
* History of major immunologic reaction (such as serum sickness or anaphylactoid reaction) to an Immunoglobulin G (IgG) containing agent (such as intravenous (IV) gamma globulin, a fusion protein, or monoclonal antibody)
* Confounders of the assessment of neurologic response including other diseases that produce chronic neurologic manifestations (such as amyotrophic lateral sclerosis, Guillain-Barre syndrome, Lyme disease, myasthenia gravis, etc.)
* Prior exposure to anti-IL-12 antibodies
* Confounders of safety assessment, such as an unstable medical condition not related to MS (including those requiring an adjustment of treatment in the four weeks prior to Screening)
* Exacerbation of asthma requiring hospitalization in the ten years prior to Screening (subjects with asthma not requiring hospitalization should be discussed with the medical monitor prior to Screening)
* Pregnant or lactating females
* The following exclusionary laboratory values at screening or baseline:

  * Hemoglobin (Hgb) <10 g/dL in females or <12 g/dL in males;
  * White blood cell (WBC) count <3 x 109/L;
  * Platelet count <100 x 109/L
  * Serum aspartate transaminase (AST) or alanine transaminase (ALT) x 3 upper limits of normal (ULN);
  * Serum total bilirubin >/= 3 mg/dL (>/= 51 x mol/L)
  * Serum creatinine >1.6 mg/dL (> 141 x mol/L)
* Subject has a recent history of substance abuse or psychiatric illness that could preclude compliance with the protocol
* In the eight weeks prior to study drug administration, the subject has received a transfusion of any blood product, or has had 500 mL or more of blood removed by repetitive or one-time blood donation, plasmapheresis, or plasma exchange, or has lost 550 mL or more blood because of hemorrhage; or
* For any reason, subject is considered by the investigator to be an unsuitable candidate to receive ABT-874.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 215 (Actual)
Dates: Start 2004-04; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Comparison of the cumulative number of Gd enhanced (T1 weighted) lesions during the treatment phase | 24 weeks
Safety and clinical laboratory parameters | monthly
vital signs | monthly

SECONDARY OUTCOMES:
Magnetic Resonance Imaging endpoints | Screening
Magnetic Resonance Imaging endpoints | Baseline (Week 0)
Magnetic Resonance Imaging endpoints | Every 4 weeks after baseline through Week 24
Magnetic Resonance Imaging endpoints | Every 12 weeks from Week 26 to Week 120
Magnetic Resonance Imaging endpoints | Early Termination

CONTACTS AND LOCATIONS:
Overall Officials: Martin Kaul, MD, Study Chair — AbbVie
Locations (44):
- United States (27):
  - Site Reference ID/Investigator# 107, Phoenix, Arizona
  - Site Reference ID/Investigator# 163, Sun City, Arizona
  - Site Reference ID/Investigator# 156, Little Rock, Arkansas
  - Site Reference ID/Investigator# 154, Irvine, California
  - Site Reference ID/Investigator# 161, Laguna Hills, California
  - Site Reference ID/Investigator# 84, Sacramento, California
  - Site Reference ID/Investigator# 119, Boulder, Colorado
  - Site Reference ID/Investigator# 111, Miami, Florida
  - Site Reference ID/Investigator# 151, Tallahassee, Florida
  - Site Reference ID/Investigator# 108, Atlanta, Georgia
  - Site Reference ID/Investigator# 109, Atlanta, Georgia
  - Site Reference ID/Investigator# 105, Northbrook, Illinois
  - Site Reference ID/Investigator# 152, Indianapolis, Indiana
  - Site Reference ID/Investigator# 258, Lenexa, Kansas
  - Site Reference ID/Investigator# 261, Lexington, Kentucky
  - Site Reference ID/Investigator# 116, Detroit, Michigan
  - Site Reference ID/Investigator# 158, Traverse City, Michigan
  - Site Reference ID/Investigator# 124, St Louis, Missouri
  - Site Reference ID/Investigator# 259, Henderson, Nevada
  - Site Reference ID/Investigator# 153, Lebanon, New Hampshire
  - Site Reference ID/Investigator# 110, Albany, New York
  - Site Reference ID/Investigator# 117, Charlotte, North Carolina
  - Site Reference ID/Investigator# 113, Columbus, Ohio
  - Site Reference ID/Investigator# 157, Dayton, Ohio
  - Site Reference ID/Investigator# 114, Allentown, Pennsylvania
  - Site Reference ID/Investigator# 128, Houston, Texas
  - Site Reference ID/Investigator# 155, Bennington, Vermont
- Canada (5):
  - Site Reference ID/Investigator# 132, Greenfield Park
  - Site Reference ID/Investigator# 130, Halifax
  - Site Reference ID/Investigator# 82, Ottawa
  - Site Reference ID/Investigator# 169, Sherbrooke
  - Site Reference ID/Investigator# 134, Vancouver
- Site Reference ID/Investigator# 149, Frankfurt, Germany
- Netherlands (4):
  - Site Reference ID/Investigator# 137, Breda
  - Site Reference ID/Investigator# 148, Nieuwegein
  - Site Reference ID/Investigator# 138, Nijmwegen
  - Site Reference ID/Investigator# 139, Sittard
- United Kingdom (7):
  - Site Reference ID/Investigator# 159, Liverpool
  - Site Reference ID/Investigator# 140, London
  - Site Reference ID/Investigator# 142, Newcastle upon Tyne
  - Site Reference ID/Investigator# 141, Nottingham
  - Site Reference ID/Investigator# 144, Oxford
  - Site Reference ID/Investigator# 143, Stoke-on-Trent
  - Site Reference ID/Investigator# 160, Whitechapel

REFERENCES:
- [Derived] Vollmer TL, Wynn DR, Alam MS, Valdes J. A phase 2, 24-week, randomized, placebo-controlled, double-blind study examining the efficacy and safety of an anti-interleukin-12 and -23 monoclonal antibody in patients with relapsing-remitting or secondary progressive multiple sclerosis. Mult Scler. 2011 Feb;17(2):181-91. doi: 10.1177/1352458510384496. Epub 2010 Dec 6. PMID 21135022